CLINICAL TRIAL: NCT06798831
Title: A Randomized, Observer-blind, Active-controlled Study to Describe the Safety of Recombinant Acellular Pertussis (aP) Vaccine When Administered to Healthy Adults Aged of 18-75 Years Old
Brief Title: Study Evaluating the Safety of a Recombinant Acellular Pertussis Vaccine in Adults
Acronym: PertaSafe
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioNet-Asia Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: APV301; BioNet-Asia.Co.,Ltd. (Other: BioNet-Asia.Co.,Ltd.)
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Pertussis Vaccine
Keywords: Recombinant Pertussis Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Boostrix (Active Comparator): Licensed tetanus toxoid, reduced diphtheria toxoid and acellular pertussis (Tdap) vaccine
  Interventions: Biological: Pertussis containing vaccine
- Recombinant acellular pertussis (aP) vaccine (Experimental): Licensed recombinant acellular pertussis (aP) vaccine (containing 5 µg of PTgen and 5 µg of FHA)
  Interventions: Biological: Pertussis containing vaccine

INTERVENTIONS:
Biological: Pertussis containing vaccine — Recombinant acellular pertussis (aP) vaccine (containing 5 µg of geneticallydetoxified pertussis toxin (PTgen),

SUMMARY:
This pivotal safety trial aims to extend the safety database for BioNet recombinant acellular pertussis (aP) vaccine (Pertagen®) in a larger population of adults and evaluate the incidence and characteristics of adverse drug reactions (ADRs), including uncommon events, to provide robust safety data. The study focuses on identifying and describing all ADRs following vaccination with BioNet recombinant acellular pertussis (aP) vaccine, ensuring the vaccine's safety is well-characterized in a large population. This study will also describe the lot-to-lot consistency between three lots of BioNet recombinant acellular pertussis (aP) vaccine across safety outcomes.

DETAILED DESCRIPTION:
This is a pivotal, multi-site, observer-blind, randomized, active-controlled vaccine trial in which 2400 healthy adults aged 18 to 75 years will be recruited at approximately 7:1 ratio from three sites in Bangkok, Thailand. As the aim of this trial is to extend the safety database for recombinant acellular pertussis (aP) vaccine in a larger population of adults, the active-controlled arm is added mainly to reduce selection and measurement bias through randomization and blinding methods.

ELIGIBILITY:
Inclusion Criteria:

* An adult participant will be eligible for inclusion if ALL of the following criteria are met at the time of screening:

  1. Aged 18 to 75 years (less than 76 years full of age) on the day of inclusion;
  2. Can provide written informed consent;
  3. Healthy, as established by pertinent medical history and physical examination;
  4. Capable of complying with the study protocol and procedures;
  5. For women with childbearing potential (i.e., urine pregnancy test will not be performed in females who have undergone sterilization, hysterectomy or who are post-menopausal.), must have a negative urine pregnancy test at enrollment.

Exclusion Criteria:

* A participant with ANY of the following criteria at study entry will not be eligible for participation:

  1. History of significant medical illness such as but not limited to immune deficiency, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic, renal, splenic or thymic functional abnormality as determined by the investigator based on medical history and physical examination. For those cases that are clinically stable, the investigator may include them as deemed per medical judgement.
  2. Breastfeeding women or female participants who intend to become pregnant during the study period;
  3. History of a severe allergic reaction to any vaccine (including its components);
  4. History of serious adverse event or neurological adverse event to any vaccination;
  5. Receipt of any investigational product or licensed vaccine within 30 days prior to enrollment (3 months for live-attenuated vaccines);
  6. Plan to receive tetanus, diphtheria or pertussis vaccine or plan to participate in other clinical trial during the study period;
  7. Having experienced physician-diagnosed pertussis within 5 year prior to enrollment;
  8. Receipt of diphtheria or tetanus or pertussis vaccine within 5 years prior to enrollment;
  9. Having any progressive or severe neurologic disorder, seizure disorder or recent history of Guillain-Barré syndrome;
  10. Medically significant cancer (except for benign or localized skin cancer, cancer in remission for ≥10 years);
  11. A known bleeding diathesis or any condition that may be associated with a prolonged bleeding time resulting in a problem with intramuscular injection;
  12. Suspected or known alcoholism and/or illicit drug abuse within the past 5 years;
  13. Administration of immunoglobulins and/or any blood products within 3 months preceding study entry or planned administration during the study period;
  14. History of receiving immunosuppressive drugs or systemic corticosteroid (>0.5 mg/kg of prednisolone or equivalent for more than 14 days) within 3 months prior to study entry;
  15. Has any active clinically significant finding or life-threatening disease that, in the opinion of the investigator, would increase the risk of the individual's having an adverse outcome by participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2399 (Actual)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and percentages of participants reporting any adverse drug reactions (ADRs) | 28 days after vaccination
  Incidence and percentages of participants reporting any adverse drug reactions (ADRs) within 28 days following a single booster dose of recombinant acellular pertussis (aP) vaccine.

SECONDARY OUTCOMES:
Incidence, severity, and percentages of participants reporting adverse events (AEs) | 28 days following vaccination
  Incidence, severity, and percentages of participants reporting adverse events (AEs) during 28 days following vaccination
Incidence, severity, and percentages of participants reporting serious adverse events (SAEs) | 28 days after vaccination
  Incidence, severity, and percentages of participants reporting serious adverse events (SAEs) during the study period.
Duration of AEs, ADRs, and SAEs | 28 days after vaccination
  Duration of AEs, ADRs, and SAEs, categorized by severity and MedDRA System Organ Class.
Categorization of ADRs by System Organ Class and Preferred Term | 28 days after vaccination
  Categorization of ADRs by System Organ Class and Preferred Term, based on MedDRA coding.

OTHER OUTCOMES:
The frequency and characteristics of AEs and ADRs | 28 days after vaccination
  The frequency and characteristics of AEs and ADRs across three lots of recombinant acellular pertussis (aP) vaccine.
Incidence and characteristics of unsolicited AEs and ADRs | 28 days after vaccination
  Incidence and characteristics of unsolicited AEs and ADRs pooled from all randomized controlled trials with aP vaccine including APV301, TDA206 TDA202, TDA207, PertaPrime and any relevant studies.

CONTACTS AND LOCATIONS:
Locations (3):
- Thailand (3):
  - Chula Clinical Research Center (Chula CRC), Bangkok, Bangkok
  - Queen Saovabha Memorial Institute, Thai Red Cross Society, Bangkok, Bangkok
  - Thai Red Cross AIDS and Infectious Diseases Research Centre, Bangkok, Bangkok

IPD SHARING:
Plan to Share IPD: No